CLINICAL TRIAL: NCT00875303
Title: Brief Primary Care Intervention Helps Parents With Discipline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PN Feb 2008
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Discipline
Keywords: Parents' plans to discipline their children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Routine primary care.
  Interventions: Behavioral: Control
- Multimedia intervention (Experimental)
  Interventions: Behavioral: Play Nicely program

INTERVENTIONS:
Behavioral: Play Nicely program — The intervention was the Play Nicely program, a multimedia educational program. Permission to demonstrate the program to multiple viewers was obtained from the copyright holder. English speaking caregivers viewed the 2nd English language edition and Spanish speaking caregivers viewed the Spanish edition. In the program, there are 16 options (20 options in the Spanish version) to respond to the hypothetical situation of witnessing a young child have hurtful behavior toward another child. Caregivers in the intervention group were instructed to view 4 of the interactive options of their choosing. On average, it takes 1 minute to view one option. Parents in the control group received routine primary care with their pediatrician.
  Arms: Multimedia intervention
Behavioral: Control — Routine primary care.
  Arms: Control

SUMMARY:
Play Nicely, is a 40 minute, interactive, media-rich, CD ROM that teaches parents, health care professionals, counselors, and child care workers/teachers the basics in aggression management for children ages 1-7. For more information about the program and to review results of previous studies, see www.playnicely.org. The objective of this study is to determine if using this brief intervention during the well child visit can affect parents' plans to discipline their children.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking parents of 1-5 year old children presenting to the Vanderbilt Primary Care Clinic for a well child visit.

Exclusion Criteria:

* Caregiver could not speak English or Spanish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
As a result of the well child visit, parents' plans to change how they discipline their children. | Same day as well child visit.

SECONDARY OUTCOMES:
Parents' report of number of minutes of discussion between physician and parent about childhood behavior or discipline. | Same day

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Pediatric Primary Care Clinic, Nashville, Tennessee, United States

REFERENCES:
- [Background] Scholer SJ, Brokish PA, Mukherjee AB, Gigante J. A violence-prevention program helps teach medical students and pediatric residents about childhood aggression. Clin Pediatr (Phila). 2008 Nov;47(9):891-900. doi: 10.1177/0009922808319965. Epub 2008 Jul 14. PMID 18626103
- [Background] Scholer SJ, Walkowski CA, Bickman L. Voluntary or required viewing of a violence prevention program in pediatric primary care. Clin Pediatr (Phila). 2008 Jun;47(5):461-8. doi: 10.1177/0009922807311731. Epub 2008 Jan 23. PMID 18216389
- [Background] Scholer SJ, Mukherjee AB, Gibbs KI, Memon S, Jongeward KL. Parents view a brief violence prevention program in clinic. Clin Pediatr (Phila). 2007 Oct;46(8):724-34. doi: 10.1177/0009922807302508. Epub 2007 Jul 19. PMID 17641130
- [Background] Scholer SJ, Cherry R, Garrard HG 4th, Gupta AO, Mace R, Greeley N. A multimedia program helps parents manage childhood aggression. Clin Pediatr (Phila). 2006 Nov;45(9):835-40. doi: 10.1177/0009922806294217. PMID 17041171
- [Background] Scholer SJ, Nix RL, Patterson B. Gaps in pediatricians' advice to parents regarding early childhood aggression. Clin Pediatr (Phila). 2006 Jan-Feb;45(1):23-8. doi: 10.1177/000992280604500104. PMID 16429212
- [Result] Scholer SJ, Hudnut-Beumler J, Dietrich MS. A brief primary care intervention helps parents develop plans to discipline. Pediatrics. 2010 Feb;125(2):e242-9. doi: 10.1542/peds.2009-0874. Epub 2010 Jan 18. PMID 20083523
- [Result] Scholer SJ, Hudnut-Beumler J, Dietrich MS. The effect of physician--parent discussions and a brief intervention on caregivers' plan to discipline: is it time for a new approach? Clin Pediatr (Phila). 2011 Aug;50(8):712-9. doi: 10.1177/0009922811400730. Epub 2011 Mar 10. PMID 21393318
- [Derived] Scholer SJ, Hudnut-Beumler J, Dietrich MS. Why parents value a brief required primary care intervention that teaches discipline strategies. Clin Pediatr (Phila). 2012 Jun;51(6):538-45. doi: 10.1177/0009922812439241. Epub 2012 Apr 11. PMID 22496174